CLINICAL TRIAL: NCT07071350
Title: Randomized Controlled Trial of Treatment to Optimize Heart Rate Variability for Persistent Post-Concussion Symptoms
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20031279
Record Dates: First submitted 2025-06-26; First posted 2025-07-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Autonomic Nervous System Disease; Concussive Injury; Mild Traumatic Brain Injury; Post Traumatic Stress Disorder; Persistent Post Concussion Syndrome
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic | interventions — Patient Health Questionnaire

STUDY DESIGN:
Intervention Model Description: This study, a randomized, controlled trial (RCT) of an easily implemented, mechanism-driven, behavioral intervention using HRV biofeedback (HRV-B) to treat PPCS among adults, including c-Vs and SMs, with history of single or repeated mTBI from blast-related or other mechanism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart rate variability biofeedback (HRV-B) (Experimental): Behavioral intervention using HRV biofeedback (HRV-B) to treat Persistent Post-Concussion Symptoms (PPCS) among adults, including Combat Veterans (c-Vs) and Service Members (SMs), with history of single or repeated mTBI from blast-related or other mechanism.
  Interventions: Other: HRV Coherence Ratio; Behavioral: NSI; Behavioral: Pittsburgh Sleep Quality Index (PSQI); Behavioral: Quantitative Sleep Measures; Behavioral: Patient Global Impression of Change (PGIC); Behavioral: Cognitive Performance/NIH Toolbox Cognitive Battery; Other: Pain Interference/TBI-QoL Pain Interference Short-Form; Behavioral: Patient Health Questionnaire-9 (PHQ-9); Behavioral: PTSD Checklist for DSM-5 (PCL-5); Other: HRV Biofeedback (HRV-B)
- Education (Experimental): Psychoeducational treatment
  Interventions: Other: HRV Coherence Ratio; Behavioral: NSI; Behavioral: Pittsburgh Sleep Quality Index (PSQI); Behavioral: Quantitative Sleep Measures; Behavioral: Patient Global Impression of Change (PGIC); Behavioral: Cognitive Performance/NIH Toolbox Cognitive Battery; Other: Pain Interference/TBI-QoL Pain Interference Short-Form; Behavioral: Patient Health Questionnaire-9 (PHQ-9); Behavioral: PTSD Checklist for DSM-5 (PCL-5); Other: Psychoeducational (Edu) Comparator Intervention

INTERVENTIONS:
Other: HRV Coherence Ratio — Evaluates autonomic function and the intervention process's efficacy, specifically resonance frequency breathing. The HRV Coherence Ratio will be quantified using a non-invasive procedure during resonance frequency breathing conditions and a standardized definition.
Behavioral: NSI — This inventory assesses the overall symptom burden, including post-concussion symptoms, on a 5-point scale. It is a well-established measure used by the Department of Defense (DoD) and VA and in mTBI outcome research at large, and includes 27 items that capture vestibular, somatosensory, cognitive, and affective symptoms.
Behavioral: Pittsburgh Sleep Quality Index (PSQI) — It includes seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Higher PSQI scores indicate poorer sleep quality.
Behavioral: Quantitative Sleep Measures — Measured using wrist actigraphy, which provides objective data on sleep parameters such as sleep latency, duration, efficiency, fragmentation, and wake time after sleep onset (WASO). Participants will wear the actigraphy monitors at baseline, post-training, and follow-up assessments.
Behavioral: Patient Global Impression of Change (PGIC) — It evaluates patients' perceptions of clinically meaningful changes in their condition following the intervention. It is considered the gold standard for such assessments.
Behavioral: Cognitive Performance/NIH Toolbox Cognitive Battery — Assessed using the NIH Toolbox Cognitive Battery, which measures executive function, episodic memory, working memory, processing speed, language, attention, and reading through a brief, computer-based test
Other: Pain Interference/TBI-QoL Pain Interference Short-Form — Evaluated using the TBI-QoL Pain Interference Short-Form, a 10-item questionnaire that measures the extent to which pain interferes with daily activities and overall quality of life. Each BPI-I item is scored from 0="Does not interfere" to 10="Completely interferes," and the scale score is the mean of the 7 items. Scores range from 0 to 10 with higher scores indicating greater pain interference.
Behavioral: Patient Health Questionnaire-9 (PHQ-9) — Assesses the severity of depressive symptoms over the past two weeks. Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Behavioral: PTSD Checklist for DSM-5 (PCL-5) — The PCL-5 (PTSD Checklist for DSM-5) is a screening tool that assesses the presence and severity of PTSD symptoms according to DSM-5 criteria. It's not a diagnostic tool itself but helps clinicians determine if further evaluation is needed. Scores range from 0 to 80, with higher scores indicating more severe symptoms.
Other: HRV Biofeedback (HRV-B) — participants will receive weekly biofeedback training over a six-week period. Each session includes approximately 30-40 minutes of biofeedback training where participants are affixed with HRV monitoring equipment. They will be guided to synchronize their heart rate variability (HRV) through slow diaphragmatic breathing and focusing on positive emotions. This process involves viewing real-time HRV patterns on a computer monitor, with coaching to help participants achieve resonant frequency breathing.
  Arms: Heart rate variability biofeedback (HRV-B)
Other: Psychoeducational (Edu) Comparator Intervention — Six weekly meetings 30-40 minutes, viewing standardized educational content on concussion recovery. No information on breathing will be provided to participants in the Edu group.
  Arms: Education

SUMMARY:
Many combat veterans (c-Vs), service members (SMs) and civilians with mild traumatic brain injury (mTBI, also termed concussion) suffer from persistent post-concussion symptoms (PPCS) that degrade physical and cognitive well-being and have been linked with early neurodegeneration. PPCS include somatosensory (e.g., headache, disturbed vision), vestibular (e.g., dizzy, clumsy), cognitive (e.g., executive function, memory) and affective symptoms (e.g., sleep disturbance, irritability, depression). A key pathological process that provokes and perpetuates PPCS is autonomic nervous system (ANS) dysfunction such as unremitting sympathetic nervous system activation that also exacerbates other pathology such as inflammation. ANS activity can be readily quantified by measuring heart rate variability (HRV), or the variation in heart rate over time, which serves as a valid index of both physiological and psychological health

DETAILED DESCRIPTION:
This study, a randomized, controlled trial (RCT) of an easily implemented, mechanism-driven, behavioral intervention using HRV biofeedback (HRV-B) to treat PPCS among adults, including c-Vs and SMs, with history of single or repeated mTBI from blast-related or other mechanism. Specifically, we study an intervention for persons with PPCS that promotes sustained functional recovery during the chronic phase of injury, which addresses psychological health and cognitive functioning, and has the potential to address neurodegenerative processes associated with TBI and treat co-occurring TBI and psychological health conditions. Importantly, the intervention is non-invasive, rapidly deployable, and is based on the pathophysiology and a theoretical mechanism of PPCS. Secondarily, this project also has the potential as a more generalized solution to increase readiness and psychological resilience in individuals, small teams, families, and communities to ameliorate the potential negative impacts of specific military and life stressors.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* History of military service
* Self-Reported hx of 1 or more mild TBI
* Most recent TBI more than 1 year ago
* Significant Persistent Post-Concussion Symptom burden (Neurobehavioral Symptom Inventory [NSI] total score greater than or equal to 20).
* Current Sleep Difficulties
* Fluent English
* Able to provide Informed Consent

Exclusion Criteria:

* Any TBI with severity greater than mild (i.e., Moderate or Severe TBI defined as initial injury loss of consciousness (LOC) duration >30 minutes, posttraumatic amnesia (PTA) duration >24 hours, or traumatic hemorrhage on head computerized tomography (CT) and determined by the study investigator based on information gathered during administration of the study's validated TBI structured interview instrument.
* Conditions or medications that can affect HRV measurement (pacemaker or an implant that stimulates your heart (e.g., cardioverter-defibrillator or ICD); heart transplant or heart surgery within the last year, including bypass or other surgery, but not including a stent)
* Hx of stroke
* Mental conditions that may impede adherence (e.g., dementia, psychotic disorder, panic disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) | Baseline to end of study procedures (11 weeks)
  The Neurobehavioral Symptom Inventory (NSI) is a 22-item self-report questionnaire used to assess the severity of neurobehavioral symptoms following traumatic brain injury (TBI), particularly postconcussion symptoms. It's a widely used tool in TBI research and clinical evaluation by the Department of Defense and Department of Veterans Affairs. The total score ranges from 0 to 88, with higher scores indicating more severe post-concussive symptoms

SECONDARY OUTCOMES:
Heart Rate Variability Biofeedback (HRV-B) | Baseline to end of study procedures (11 weeks)
  It is a biofeedback technique that trains individuals to regulate their heart rate variability (HRV) through breathing exercises. It aims to improve self-regulation, reduce stress, and enhance overall well-being by strengthening the parasympathetic nervous system. HRV varies depending on age, fitness level, and overall health, and falls between 60 and 100 ms for most individuals. However, it is important to note that a "good" HRV may differ from person to person based on their individual circumstances.
NIH Toolbox Cognitive Battery | Baseline to end of study procedures (11 weeks)
  Assessed using the NIH Toolbox Cognitive Battery, which measures executive function, episodic memory, working memory, processing speed, language, attention, and reading through a brief, computer-based test
TBI-QoL Pain Interference Short-Form | Baseline to end of study procedures (11 weeks)
  Evaluated using the TBI-QoL Pain Interference Short-Form, a 10-item questionnaire that measures the extent to which pain interferes with daily activities and overall quality of life. Each BPI-I item is scored from 0="Does not interfere" to 10="Completely interferes," and the scale score is the mean of the 7 items. Scores range from 0 to 10 with higher scores indicating greater pain interference.
Patient Health Questionnaire-9 (PHQ-9) | Baseline to end of study procedures (11 weeks)
  Patient Health Questionnaire-9 (PHQ-9) Assesses the severity of depressive symptoms over the past two weeks. Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression
PCL-5 (PTSD Checklist for DSM-5) | Baseline to end of study procedures (11 weeks)
  The PCL-5 (PTSD Checklist for DSM-5) is a screening tool that assesses the presence and severity of PTSD symptoms according to DSM-5 criteria. It's not a diagnostic tool itself but helps clinicians determine if further evaluation is needed. Scores range from 0 to 80, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: James Burch, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No